CLINICAL TRIAL: NCT04143061
Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Healthy Adults, Adolescents, Children, and Toddlers in India and Healthy Adolescents and Children in the Republic of South Africa
Acronym: MET55
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MET55; U1111-1183-6581 (Registry Identifier: ICTRP); MET55 (Other: Sanofi Identifier); 2020-004341-36 (EudraCT Number)
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Meningococcal Immunization; Healthy Volunteers
MeSH Terms: interventions — Meningococcal Vaccines; Vaccines

STUDY DESIGN:
Intervention Model Description: Toddlers (open-label), children, adolescents and adults aged 12 months and above are enrolled in India, and children and adolescents aged 2 to 17 years are included in RSA. The older populations (adults) are recruited before initiating the study in children and adolescents younger than 17 years of age in India.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial is a modified double-blind trial (except for toddlers in India), which means that the participant's parent / legally acceptable representative, the Investigator, and other study personnel remain unaware of the treatment assignments throughout the trial. An unblinded vaccine administrator administer the appropriate vaccine but is not involved in safety data collection. The Sponsor and laboratory personnel performing the serology testing are also blinded to treatment assignments throughout the trial until database lock.
  It will be open-label for toddlers population in India.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Group 1 (Experimental): MenACYW conjugate vaccine, 1 vaccination, adults in India aged 18 to 55 years
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid conjugate vaccine
- Group 2 (Active Comparator): Menactra® conjugate vaccine, 1 vaccination, adults in India aged 18 to 55 years
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W-135) diphtheria toxoid conjugate vaccine
- Group 3 (Experimental): MenACYW conjugate vaccine, 1 vaccination, adults in India aged ≥ 56 years
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid conjugate vaccine
- Group 4 (Active Comparator): Quadri Meningo™, 1 vaccination, adults in India aged ≥ 56 years
  Interventions: Biological: Meningococcal polysaccharide (serogroups A, C, Y and W-135) vaccine
- Group 5 (Experimental): MenACYW conjugate vaccine, 1 vaccination, children and adolescents in India aged 2 to 17 years
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid conjugate vaccine
- Group 6 (Active Comparator): Menactra®, 1 vaccination, children and adolescents in India aged 2 to 17 years
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W-135) diphtheria toxoid conjugate vaccine
- Group 7 (Experimental): MenACYW conjugate vaccine, 1 vaccination, children and adolescents in RSA aged 2 to 17 years
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid conjugate vaccine
- Group 8 (Active Comparator): Menactra®, 1 vaccination, children and adolescents in RSA aged 2 to 17 years
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W-135) diphtheria toxoid conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid conjugate vaccine — Pharmaceutical form: solution for injection; Route of administration: intramuscular, 0.5 mL
  Other Names: MenACYW conjugate vaccine
  Arms: Group 1; Group 3; Group 5; Group 7
Biological: Meningococcal polysaccharide (serogroups A,C,Y and W-135) diphtheria toxoid conjugate vaccine — Pharmaceutical form: sterile aqueous solution; Route of administration: intramuscular, 0.5 mL
  Other Names: Menactra®
  Arms: Group 2; Group 6; Group 8
Biological: Meningococcal polysaccharide (serogroups A, C, Y and W-135) vaccine — Pharmaceutical form: reconstituted solution for injection; Route of administration: intramuscular, 0.5 mL
  Other Names: Quadri Meningo™
  Arms: Group 4

SUMMARY:
This will be a Phase III, modified double-blind (open-label for toddlers in India), randomized, parallel-group, active-controlled, step-wise, multi-center study to compare and describe the immunogenicity and safety of MenACYW conjugate vaccine when administered as a single dose in healthy adults, adolescents, children, and toddlers in India and a modified double-blind, randomized, parallel-group, active-controlled, multi-center study to compare and describe the immunogenicity and safety of MenACYW conjugate vaccine when administered as a single dose in healthy adolescents and children in RSA.

DETAILED DESCRIPTION:
Study duration per participant is approximately 31 to 45 days

ELIGIBILITY:
Inclusion Criteria:

- Age in the defined range on the day of inclusion: For Adults: Aged ≥ 18 years on the day of inclusion For Children and Adolescents: Aged 2 to 17 years on the day of inclusion For Toddlers: Aged 12 to 23 months† on the day of inclusion

- Z-score of ≥ -2 standard deviations (SD) on the Weight-for-height table of the World Health Organization (WHO) Child Growth Standards: For toddlers and children: Toddlers aged 12 to 23 months and Children aged 2 to 5 years had a Z-score of ≥ -2 SD on the Weight-for-height table of the WHO Child Growth Standards

* Informed consent obtained For adults: Informed consent form has been signed and dated by the subject and by an independent witness, if required by local regulations For toddlers, children, and adolescents: Assent form has been signed and dated by the subject (for subjects 7 to 17 years of age), and informed consent form has been signed and dated by the parent(s) or legally acceptable representative and by an independent witness, if required by local regulations
* Were able to attend all scheduled visits and to comply with all trial procedures For adults: Were able to attend all scheduled visits and to comply with all trial procedures For toddlers, children, and adolescents: Participants and parent / legally acceptable representative were able to attend all scheduled visits and to comply with all trial procedures
* For Toddlers: All toddlers were due to receive an age-recommended RPV on D0

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential and was not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche, or post-menopausal for at least 1 year, or surgically sterile
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks (28 days) preceding the IMP or planned receipt of any vaccine in the 4 weeks following vaccination except for oral poliovirus vaccine (OPV) in India, received during national immunization days. In India, OPV might have been received with a gap of at least 2 weeks before the IMP. This exception included monovalent and bivalent OPV.
* Previous vaccination against meningococcal disease with either the IMP or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B serogroup containing vaccine)
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically
* At high risk for meningococcal infection during the trial (specifically, but not limited to, subjects with persistent complement deficiency, with anatomic or functional asplenia, or subjects traveling to countries with high endemic or epidemic disease)
* Known systemic hypersensitivity to latex or to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Verbal report of thrombocytopenia, as reported by the subject or the subject's parent / legally acceptable representative, contraindicating intramuscular vaccination in the Investigator's opinion
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion
* Personal history of Guillain-Barré syndrome
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine within 10 years of the proposed study vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion
* Any condition which, in the opinion of the Investigator, might have interfered with the evaluation of the study objectives.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination, febrile illness (temperature ≥ 38.0°C), persistent diarrhea, vomiting. A prospective subject was not included in the study until the condition has been resolved or the febrile event has been subsided
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1328 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (17):
- India (10):
  - Investigational Site Number : 3560002, Bangalore
  - Investigational Site Number : 3560016, Belagavi
  - Investigational Site Number : 3560007, Chennai
  - Investigational Site Number : 3560004, Hyderabad
  - Investigational Site Number : 3560011, Kolkata
  - Investigational Site Number : 3560012, Mysore
  - Investigational Site Number : 3560015, Odisha
  - Investigational Site Number : 3560003, Pune
  - Investigational Site Number : 3560008, Pune
  - Investigational Site Number : 3560010, Punjab
- South Africa (7):
  - Investigational Site Number : 7100004, Bertsham
  - Investigational Site Number : 7100007, Bloemfontein
  - Investigational Site Number : 7100005, Cape Town
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100001, Middelburg
  - Investigational Site Number : 7100006, Pretoria
  - Investigational Site Number : 7100003, Soweto

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 17 investigational sites: 10 centers in India and 7 centers in the Republic of South Africa (RSA) between 30 December 2019 and 28 January 2023.
Pre-assignment Details: A total of 1328 participants were enrolled and randomized in the study. Toddlers were not enrolled in this study.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Adult participants aged 18 to 55 years in India received a single dose of 0.5 milliliter (mL) meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid conjugate vaccine [MenACYW conjugate vaccine] as an intramuscular (IM) injection on Day 0.
- Group 2: Menactra®: Adult participants aged 18 to 55 years in India received a single dose of 0.5 mL meningococcal (groups A, C, Y and W-135) polysaccharide diphtheria toxoid conjugate vaccine [Menactra®] as an IM injection on Day 0.
- Group 3: MenACYW Conjugate Vaccine: Adult participants aged ≥56 years in India received a single dose of 0.5 mL MenACYW conjugate vaccine as an IM injection on Day 0.
- Group 4: Quadri Meningo™/Locally Available Licensed Meningococcal Vaccine: Adult participants aged ≥56 years in India received a single dose of 0.5 mL meningococcal polysaccharide vaccine (group A, C, Y and W135) [Quadri Meningo™] or any locally available licensed meningococcal vaccine as an IM injection on Day 0.
- Group 5: MenACYW Conjugate Vaccine: Children and adolescent participants aged 2 to 17 years in India received a single dose of 0.5 mL MenACYW conjugate vaccine as an IM injection on Day 0.
- Group 6: Menactra®: Children and adolescent participants aged 2 to 17 years in India received a single dose of 0.5 mL Menactra® as an IM injection on Day 0.
- Group 7: MenACYW Conjugate Vaccine: Children and adolescent participants aged 2 to 17 years in RSA received a single dose of 0.5 mL MenACYW conjugate vaccine as an IM injection on Day 0.
- Group 8: Menactra®: Children and adolescent participants aged 2 to 17 years in RSA received a single dose of 0.5 mL Menactra® as an IM injection on Day 0.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® | Group 3: MenACYW Conjugate Vaccine | Group 4: Quadri Meningo™/Locally Available Licensed Meningococcal Vaccine | Group 5: MenACYW Conjugate Vaccine | Group 6: Menactra® | Group 7: MenACYW Conjugate Vaccine | Group 8: Menactra®
Started | 98 | 100 | 100 | 100 | 232 | 233 | 233 | 232
Completed | 96 | 100 | 100 | 100 | 224 | 229 | 226 | 220
Not Completed | 2 | 0 | 0 | 0 | 8 | 4 | 7 | 12
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 8 | 3 | 2 | 7

BASELINE CHARACTERISTICS:
Population: Randomized study participants included all enrolled participants for whom an injection group had been allocated and who had any available data in case report form.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Adult participants aged 18 to 55 years in India received a single dose of 0.5 mL MenACYW conjugate vaccine as an IM injection on Day 0.
- Group 2: Menactra®: Adult participants aged 18 to 55 years in India received a single dose of 0.5 mL Menactra® as an IM injection on Day 0.
- Group 4: Quadri Meningo™/Locally Available Licensed Meningococcal Vaccine: Adult participants aged ≥56 years in India received a single dose of 0.5 mL Quadri Meningo™ or any locally available licensed meningococcal vaccine as an IM injection on Day 0.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® | Group 3: MenACYW Conjugate Vaccine | Group 4: Quadri Meningo™/Locally Available Licensed Meningococcal Vaccine | Group 5: MenACYW Conjugate Vaccine | Group 6: Menactra® | Group 7: MenACYW Conjugate Vaccine | Group 8: Menactra® | Total
Number analyzed (Participants) | 98 | 100 | 100 | 100 | 232 | 233 | 233 | 232 | 1328
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (9.21) | 34.8 (9.05) | 61.7 (6.09) | 61.1 (5.61) | 9.39 (4.19) | 9.34 (4.10) | 9.45 (4.01) | 9.19 (4.19) | 21.1 (20.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 24 | 31 | 101 | 118 | 123 | 110 | 568
  Male | 68 | 69 | 76 | 69 | 131 | 115 | 110 | 122 | 760
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 98 | 100 | 100 | 100 | 232 | 233 | 0 | 0 | 863
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 142 | 139 | 281
  White | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 10 | 19
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 9
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 15
  Mixed Origin | 0 | 0 | 0 | 0 | 0 | 0 | 70 | 71 | 141

OUTCOME MEASURES:

1. Primary Outcome: Group 5 + 7 and Group 6 + 8: Percentage of Participants Who Achieved Antibody Titers ≥1:8 Against Meningococcal Serogroups A, C, Y, and W
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured by serum bactericidal assay using human complement (hSBA). Percentages are rounded off to the tenth decimal place. As pre-specified in protocol, the endpoint was assessed in children and adolescents aged 2 to 17 years in India and RSA as combined groups: Group 5 + Group 7 and Group 6 + Group 8 as they received the same dose of MenACYW conjugate vaccine and Menactra® respectively.
Time Frame: Day 30 (30 days post-vaccination on Day 0)
Population: Analysis was performed on the per-protocol analysis set (PPAS) which was a subset of the full analysis set (FAS). The FAS was the subset of randomized participants who received at least 1 dose of the study vaccine and had a valid post-vaccination blood sample result. Only participants with data collected for each specific serogroup are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 5 + Group 7: MenACYW Conjugate Vaccine: Children and adolescent participants aged 2 to 17 years in India and RSA received a single dose of 0.5 mL MenACYW conjugate vaccine as an IM injection on Day 0.
- Group 6 + Group 8: Menactra®: Children and adolescent participants aged 2 to 17 years in India and RSA received a single dose of 0.5 mL Menactra® as an IM injection on Day 0.
Arm/Group | Group 5 + Group 7: MenACYW Conjugate Vaccine | Group 6 + Group 8: Menactra®
Number analyzed (Participants) | 445 | 445
percentage of participants
  Serogroup A: number analyzed (Participants) | 443 | 443
  Serogroup A | 89.6 [86.4 to 92.3] | 83.1 [79.2 to 86.4]
  Serogroup C: number analyzed (Participants) | 445 | 443
  Serogroup C | 99.3 [98.0 to 99.9] | 77.7 [73.5 to 81.4]
  Serogroup Y: number analyzed (Participants) | 445 | 443
  Serogroup Y | 96.6 [94.5 to 98.1] | 85.6 [81.9 to 88.7]
  Serogroup W | 98.7 [97.1 to 99.5] | 87.6 [84.2 to 90.6]
Statistical Analysis 1: Comparison: Group 5 + Group 7: MenACYW Conjugate Vaccine vs Group 6 + Group 8: Menactra®; Statistical analysis for Serogroup A; Test type: Non-Inferiority — The overall non-inferiority was demonstrated if the lower limit of the 2-sided 95% confidence interval (CI) was >-10% for all 4 serogroups. 95% CI of the difference was calculated from the Wilson Score method without continuity correction; Difference in percentage of participants = 6.55, 95% CI 2-sided [2.03 to 11.08]
Statistical Analysis 2: Comparison: Group 5 + Group 7: MenACYW Conjugate Vaccine vs Group 6 + Group 8: Menactra®; Statistical analysis for Serogroup C; Test type: Non-Inferiority — The overall non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >-10% for all 4 serogroups. 95% CI of the difference was calculated from the Wilson Score method without continuity correction; Difference in percentage of participants = 21.67, 95% CI 2-sided [17.82 to 25.80]
Statistical Analysis 3: Comparison: Group 5 + Group 7: MenACYW Conjugate Vaccine vs Group 6 + Group 8: Menactra®; Statistical analysis for Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 11.08, 95% CI 2-sided [7.43 to 14.89]
Statistical Analysis 4: Comparison: Group 5 + Group 7: MenACYW Conjugate Vaccine vs Group 6 + Group 8: Menactra®; Statistical analysis for Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 11.01, 95% CI 2-sided [7.86 to 14.47]

2. Secondary Outcome: Group 1 and Group 2: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured by hSBA and serum bactericidal assay using baby rabbit complement (rSBA).
Time Frame: Day 0 (pre-vaccination) and Day 30 (30 days post-vaccination on Day 0)
Population: Analysis was performed on the PPAS which was a subset of the FAS. The FAS was the subset of randomized participants who received at least 1 dose of the study vaccine and had a valid post-vaccination blood sample result. Only participants with data collected for each specific serogroup at specified timepoints are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra®
Number analyzed (Participants) | 95 | 99
titer
  hSBA: Serogroup A: Day 0 | 7.28 [6.03 to 8.78] | 9.60 [7.68 to 12.0]
  hSBA: Serogroup A: Day 30: number analyzed (Participants) | 94 | 99
  hSBA: Serogroup A: Day 30 | 52.8 [34.7 to 80.3] | 39.2 [27.8 to 55.3]
  hSBA: Serogroup C: Day 0 | 6.20 [4.99 to 7.70] | 7.05 [5.53 to 8.99]
  hSBA: Serogroup C: Day 30 | 551 [365 to 831] | 107 [68.8 to 165]
  hSBA: Serogroup Y: Day 0 | 5.24 [3.86 to 7.11] | 4.03 [3.09 to 5.25]
  hSBA: Serogroup Y: Day 30 | 119 [80.2 to 177] | 47.4 [30.7 to 73.1]
  hSBA: Serogroup W: Day 0 | 4.18 [3.39 to 5.15] | 4.17 [3.39 to 5.14]
  hSBA: Serogroup W: Day 30: number analyzed (Participants) | 94 | 99
  hSBA: Serogroup W: Day 30 | 106 [72.8 to 153] | 63.1 [44.7 to 89.1]
  rSBA: Serogroup A: Day 0: number analyzed (Participants) | 45 | 47
  rSBA: Serogroup A: Day 0 | 194 [81.3 to 463] | 64.0 [25.9 to 158]
  rSBA: Serogroup A: Day 30: number analyzed (Participants) | 45 | 48
  rSBA: Serogroup A: Day 30 | 10644 [7745 to 14629] | 4467 [3428 to 5820]
  rSBA: Serogroup C: Day 0: number analyzed (Participants) | 45 | 49
  rSBA: Serogroup C: Day 0 | 5.88 [3.51 to 9.86] | 4.88 [3.00 to 7.93]
  rSBA: Serogroup C: Day 30: number analyzed (Participants) | 45 | 48
  rSBA: Serogroup C: Day 30 | 12227 [7923 to 18868] | 1149 [612 to 2158]
  rSBA: Serogroup Y: Day 0: number analyzed (Participants) | 44 | 43
  rSBA: Serogroup Y: Day 0 | 9.36 [4.33 to 20.2] | 9.40 [4.12 to 21.5]
  rSBA: Serogroup Y: Day 30: number analyzed (Participants) | 43 | 47
  rSBA: Serogroup Y: Day 30 | 5934 [3758 to 9372] | 3534 [2545 to 4909]
  rSBA: Serogroup W: Day 0: number analyzed (Participants) | 45 | 49
  rSBA: Serogroup W: Day 0 | 15.5 [6.49 to 37.1] | 7.56 [3.49 to 16.4]
  rSBA: Serogroup W: Day 30: number analyzed (Participants) | 45 | 48
  rSBA: Serogroup W: Day 30 | 16638 [10325 to 26812] | 7732 [4098 to 14589]

3. Secondary Outcome: Group 1 and Group 2: Percentage of Participants Who Achieved Antibody Titers ≥Pre-defined Thresholds Against Meningococcal Serogroups A, C, Y, and W
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured by hSBA and rSBA. Percentages are rounded off to the tenth decimal place. Percentage of participants who achieved antibody titers ≥1:4 and ≥1:8 by hSBA and ≥1:8 and ≥1:128 by rSBA are reported.
Time Frame: Day 0 (pre-vaccination) and Day 30 (30 days post-vaccination on Day 0)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra®
Number analyzed (Participants) | 95 | 99
percentage of participants
  hSBA: Serogroup A: Day 0: ≥1:4 | 81.1 [71.7 to 88.4] | 87.9 [79.8 to 93.6]
  hSBA: Serogroup A: Day 0: ≥1:8 | 61.1 [50.5 to 70.9] | 72.7 [62.9 to 81.2]
  hSBA: Serogroup A: Day 30: ≥1:4: number analyzed (Participants) | 94 | 99
  hSBA: Serogroup A: Day 30: ≥1:4 | 87.2 [78.8 to 93.2] | 93.9 [87.3 to 97.7]
  hSBA: Serogroup A: Day 30: ≥1:8: number analyzed (Participants) | 94 | 99
  hSBA: Serogroup A: Day 30: ≥1:8 | 76.6 [66.7 to 84.7] | 87.9 [79.8 to 93.6]
  hSBA: Serogroup C: Day 0: ≥1:4 | 69.5 [59.2 to 78.5] | 69.7 [59.6 to 78.5]
  hSBA: Serogroup C: Day 0: ≥1:8 | 47.4 [37.0 to 57.9] | 50.5 [40.3 to 60.7]
  hSBA: Serogroup C: Day 30: ≥1:4 | 98.9 [94.3 to 100] | 93.9 [87.3 to 97.7]
  hSBA: Serogroup C: Day 30: ≥1:8 | 96.8 [91.0 to 99.3] | 88.9 [81.0 to 94.3]
  hSBA: Serogroup Y: Day 0: ≥1:4 | 38.9 [29.1 to 49.5] | 30.3 [21.5 to 40.4]
  hSBA: Serogroup Y: Day 0: ≥1:8 | 29.5 [20.6 to 39.7] | 24.2 [16.2 to 33.9]
  hSBA: Serogroup Y: Day 30: ≥1:4 | 93.7 [86.8 to 97.6] | 82.8 [73.9 to 89.7]
  hSBA: Serogroup Y: Day 30: ≥1:8 | 92.6 [85.4 to 97.0] | 76.8 [67.2 to 84.7]
  hSBA: Serogroup W: Day 0: ≥1:4 | 44.2 [34.0 to 54.8] | 44.4 [34.5 to 54.8]
  hSBA: Serogroup W: Day 0: ≥1:8 | 29.5 [20.6 to 39.7] | 29.3 [20.6 to 39.3]
  hSBA: Serogroup W: Day 30: ≥1:4: number analyzed (Participants) | 94 | 99
  hSBA: Serogroup W: Day 30: ≥1:4 | 96.8 [91.0 to 99.3] | 96.0 [90.0 to 98.9]
  hSBA: Serogroup W: Day 30: ≥1:8: number analyzed (Participants) | 94 | 99
  hSBA: Serogroup W: Day 30: ≥1:8 | 93.6 [86.6 to 97.6] | 90.9 [83.4 to 95.8]
  rSBA: Serogroup A: Day 0: ≥1:8: number analyzed (Participants) | 45 | 47
  rSBA: Serogroup A: Day 0: ≥1:8 | 75.6 [60.5 to 87.1] | 61.7 [46.4 to 75.5]
  rSBA: Serogroup A: Day 0: ≥1:128: number analyzed (Participants) | 45 | 47
  rSBA: Serogroup A: Day 0: ≥1:128 | 62.2 [46.5 to 76.2] | 48.9 [34.1 to 63.9]
  rSBA: Serogroup A: Day 30: ≥1:8: number analyzed (Participants) | 45 | 48
  rSBA: Serogroup A: Day 30: ≥1:8 | 100 [92.1 to 100] | 100 [92.6 to 100]
  rSBA: Serogroup A: Day 30: ≥1:128: number analyzed (Participants) | 45 | 48
  rSBA: Serogroup A: Day 30: ≥1:128 | 100 [92.1 to 100] | 100 [92.6 to 100]
  rSBA: Serogroup C: Day 0: ≥1:8: number analyzed (Participants) | 45 | 49
  rSBA: Serogroup C: Day 0: ≥1:8 | 28.9 [16.4 to 44.3] | 24.5 [13.3 to 38.9]
  rSBA: Serogroup C: Day 0: ≥1:128: number analyzed (Participants) | 45 | 49
  rSBA: Serogroup C: Day 0: ≥1:128 | 11.1 [3.7 to 24.1] | 10.2 [3.4 to 22.2]
  rSBA: Serogroup C: Day 30: ≥1:8: number analyzed (Participants) | 45 | 48
  rSBA: Serogroup C: Day 30: ≥1:8 | 100 [92.1 to 100] | 95.8 [85.7 to 99.5]
  rSBA: Serogroup C: Day 30: ≥1:128: number analyzed (Participants) | 45 | 48
  rSBA: Serogroup C: Day 30: ≥1:128 | 100 [92.1 to 100] | 89.6 [77.3 to 96.5]
  rSBA: Serogroup Y: Day 0: ≥1:8: number analyzed (Participants) | 44 | 43
  rSBA: Serogroup Y: Day 0: ≥1:8 | 29.5 [16.8 to 45.2] | 25.6 [13.5 to 41.2]
  rSBA: Serogroup Y: Day 0: ≥1:128: number analyzed (Participants) | 44 | 43
  rSBA: Serogroup Y: Day 0: ≥1:128 | 25.0 [13.2 to 40.3] | 23.3 [11.8 to 38.6]
  rSBA: Serogroup Y: Day 30: ≥1:8: number analyzed (Participants) | 43 | 47
  rSBA: Serogroup Y: Day 30: ≥1:8 | 97.7 [87.7 to 99.9] | 100 [92.5 to 100]
  rSBA: Serogroup Y: Day 30: ≥1:128: number analyzed (Participants) | 43 | 47
  rSBA: Serogroup Y: Day 30: ≥1:128 | 97.7 [87.7 to 99.9] | 100 [92.5 to 100]
  rSBA: Serogroup W: Day 0: ≥1:8: number analyzed (Participants) | 45 | 49
  rSBA: Serogroup W: Day 0: ≥1:8 | 35.6 [21.9 to 51.2] | 20.4 [10.2 to 34.3]
  rSBA: Serogroup W: Day 0: ≥1:128: number analyzed (Participants) | 45 | 49
  rSBA: Serogroup W: Day 0: ≥1:128 | 31.1 [18.2 to 46.6] | 20.4 [10.2 to 34.3]
  rSBA: Serogroup W: Day 30: ≥1:8: number analyzed (Participants) | 45 | 48
  rSBA: Serogroup W: Day 30: ≥1:8 | 100 [92.1 to 100] | 97.9 [88.9 to 99.9]
  rSBA: Serogroup W: Day 30: ≥1:128: number analyzed (Participants) | 45 | 48
  rSBA: Serogroup W: Day 30: ≥1:128 | 100 [92.1 to 100] | 97.9 [88.9 to 99.9]

4. Secondary Outcome: Group 3 and Group 4: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured by hSBA and rSBA.
Time Frame: Day 0 (pre-vaccination) and Day 30 (30 days post-vaccination on Day 0)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 3: MenACYW Conjugate Vaccine | Group 4: Quadri Meningo™/Locally Available Licensed Meningococcal Vaccine
Number analyzed (Participants) | 97 | 96
titer
  hSBA: Serogroup A: Day 0 | 15.3 [12.2 to 19.3] | 12.5 [10.2 to 15.4]
  hSBA: Serogroup A: Day 30: number analyzed (Participants) | 96 | 96
  hSBA: Serogroup A: Day 30 | 56.6 [38.2 to 83.9] | 36.2 [26.8 to 48.8]
  hSBA: Serogroup C: Day 0 | 8.00 [6.18 to 10.4] | 8.00 [6.13 to 10.4]
  hSBA: Serogroup C: Day 30 | 393 [255 to 606] | 159 [102 to 248]
  hSBA: Serogroup Y: Day 0 | 6.36 [4.57 to 8.86] | 6.97 [5.03 to 9.68]
  hSBA: Serogroup Y: Day 30 | 197 [127 to 303] | 55.4 [35.5 to 86.4]
  hSBA: Serogroup W: Day 0 | 4.42 [3.53 to 5.54] | 5.66 [4.40 to 7.27]
  hSBA: Serogroup W: Day 30 | 90.8 [60.4 to 137] | 34.6 [23.5 to 51.2]
  rSBA: Serogroup A: Day 0: number analyzed (Participants) | 48 | 47
  rSBA: Serogroup A: Day 0 | 83.0 [37.0 to 186] | 46.3 [20.1 to 106]
  rSBA: Serogroup A: Day 30: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup A: Day 30 | 5834 [3730 to 9124] | 4677 [2935 to 7455]
  rSBA: Serogroup C: Day 0: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup C: Day 0 | 6.47 [3.69 to 11.3] | 5.53 [3.06 to 9.99]
  rSBA: Serogroup C: Day 30: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup C: Day 30 | 9304 [5532 to 15649] | 3283 [1680 to 6415]
  rSBA: Serogroup Y: Day 0: number analyzed (Participants) | 45 | 46
  rSBA: Serogroup Y: Day 0 | 6.86 [3.33 to 14.1] | 8.24 [3.94 to 17.3]
  rSBA: Serogroup Y: Day 30: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup Y: Day 30 | 4274 [2640 to 6917] | 1119 [529 to 2366]
  rSBA: Serogroup W: Day 0: number analyzed (Participants) | 48 | 46
  rSBA: Serogroup W: Day 0 | 11.6 [5.55 to 24.4] | 12.4 [5.04 to 30.4]
  rSBA: Serogroup W: Day 30: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup W: Day 30 | 6626 [3243 to 13539] | 2304 [925 to 5739]

5. Secondary Outcome: Group 3 and Group 4: Percentage of Participants Who Achieved Antibody Titers ≥Pre-defined Thresholds Against Meningococcal Serogroups A, C, Y, and W
Description: as for outcome 3
Time Frame: Day 0 (pre-vaccination) and Day 30 (30 days post-vaccination on Day 0)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine | Group 4: Quadri Meningo™/Locally Available Licensed Meningococcal Vaccine
Number analyzed (Participants) | 97 | 96
percentage of participants
  hSBA: Serogroup A: Day 0: ≥1:4 | 94.8 [88.4 to 98.3] | 93.8 [86.9 to 97.7]
  hSBA: Serogroup A: Day 0: ≥1:8 | 82.5 [73.4 to 89.4] | 77.1 [67.4 to 85.0]
  hSBA: Serogroup A: Day 30: ≥1:4: number analyzed (Participants) | 96 | 96
  hSBA: Serogroup A: Day 30: ≥1:4 | 89.6 [81.7 to 94.9] | 96.9 [91.1 to 99.4]
  hSBA: Serogroup A: Day 30: ≥1:8: number analyzed (Participants) | 96 | 96
  hSBA: Serogroup A: Day 30: ≥1:8 | 82.3 [73.2 to 89.3] | 86.5 [78.0 to 92.6]
  hSBA: Serogroup C: Day 0: ≥1:4 | 71.1 [61.0 to 79.9] | 75.0 [65.1 to 83.3]
  hSBA: Serogroup C: Day 0: ≥1:8 | 53.6 [43.2 to 63.8] | 50.0 [39.6 to 60.4]
  hSBA: Serogroup C: Day 30: ≥1:4 | 97.9 [92.7 to 99.7] | 92.7 [85.6 to 97.0]
  hSBA: Serogroup C: Day 30: ≥1:8 | 95.9 [89.8 to 98.9] | 89.6 [81.7 to 94.9]
  hSBA: Serogroup Y: Day 0: ≥1:4 | 45.4 [35.2 to 55.8] | 51.0 [40.6 to 61.4]
  hSBA: Serogroup Y: Day 0: ≥1:8 | 36.1 [26.6 to 46.5] | 40.6 [30.7 to 51.1]
  hSBA: Serogroup Y: Day 30: ≥1:4 | 93.8 [87.0 to 97.7] | 83.3 [74.4 to 90.2]
  hSBA: Serogroup Y: Day 30: ≥1:8 | 93.8 [87.0 to 97.7] | 79.2 [69.7 to 86.8]
  hSBA: Serogroup W: Day 0: ≥1:4 | 45.4 [35.2 to 55.8] | 54.2 [43.7 to 64.4]
  hSBA: Serogroup W: Day 0: ≥1:8 | 30.9 [21.9 to 41.1] | 38.5 [28.8 to 49.0]
  hSBA: Serogroup W: Day 30: ≥1:4 | 91.8 [84.4 to 96.4] | 90.6 [82.9 to 95.6]
  hSBA: Serogroup W: Day 30: ≥1:8 | 89.7 [81.9 to 94.9] | 79.2 [69.7 to 86.8]
  rSBA: Serogroup A: Day 0: ≥1:8: number analyzed (Participants) | 48 | 47
  rSBA: Serogroup A: Day 0: ≥1:8 | 68.8 [53.7 to 81.3] | 55.3 [40.1 to 69.8]
  rSBA: Serogroup A: Day 0: ≥1:128: number analyzed (Participants) | 48 | 47
  rSBA: Serogroup A: Day 0: ≥1:128 | 56.3 [41.2 to 70.5] | 46.8 [32.1 to 61.9]
  rSBA: Serogroup A: Day 30: ≥1:8: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup A: Day 30: ≥1:8 | 98.0 [89.1 to 99.9] | 100 [92.5 to 100]
  rSBA: Serogroup A: Day 30: ≥1:128: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup A: Day 30: ≥1:128 | 98.0 [89.1 to 99.9] | 97.9 [88.7 to 99.9]
  rSBA: Serogroup C: Day 0: ≥1:8: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup C: Day 0: ≥1:8 | 30.6 [18.3 to 45.4] | 21.3 [10.7 to 35.7]
  rSBA: Serogroup C: Day 0: ≥1:128: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup C: Day 0: ≥1:128 | 16.3 [7.3 to 29.7] | 10.6 [3.5 to 23.1]
  rSBA: Serogroup C: Day 30: ≥1:8: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup C: Day 30: ≥1:8 | 98.0 [89.1 to 99.9] | 93.6 [82.5 to 98.7]
  rSBA: Serogroup C: Day 30: ≥1:128: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup C: Day 30: ≥1:128 | 98.0 [89.1 to 99.9] | 93.6 [82.5 to 98.7]
  rSBA: Serogroup Y: Day 0: ≥1:8: number analyzed (Participants) | 45 | 46
  rSBA: Serogroup Y: Day 0: ≥1:8 | 20.0 [9.6 to 34.6] | 26.1 [14.3 to 41.1]
  rSBA: Serogroup Y: Day 0: ≥1:128: number analyzed (Participants) | 45 | 46
  rSBA: Serogroup Y: Day 0: ≥1:128 | 20.0 [9.6 to 34.6] | 21.7 [10.9 to 36.4]
  rSBA: Serogroup Y: Day 30: ≥1:8: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup Y: Day 30: ≥1:8 | 98.0 [89.1 to 99.9] | 89.4 [76.9 to 96.5]
  rSBA: Serogroup Y: Day 30: ≥1:128: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup Y: Day 30: ≥1:128 | 98.0 [89.1 to 99.9] | 89.4 [76.9 to 96.5]
  rSBA: Serogroup W: Day 0: ≥1:8: number analyzed (Participants) | 48 | 46
  rSBA: Serogroup W: Day 0: ≥1:8 | 33.3 [20.4 to 48.4] | 30.4 [17.7 to 45.8]
  rSBA: Serogroup W: Day 0: ≥1:128: number analyzed (Participants) | 48 | 46
  rSBA: Serogroup W: Day 0: ≥1:128 | 31.3 [18.7 to 46.3] | 28.3 [16.0 to 43.5]
  rSBA: Serogroup W: Day 30: ≥1:8: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup W: Day 30: ≥1:8 | 95.9 [86.0 to 99.5] | 89.4 [76.9 to 96.5]
  rSBA: Serogroup W: Day 30: ≥1:128: number analyzed (Participants) | 49 | 47
  rSBA: Serogroup W: Day 30: ≥1:128 | 93.9 [83.1 to 98.7] | 87.2 [74.3 to 95.2]

6. Secondary Outcome: Group 5 + 7 and Group 6 + 8: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured by hSBA and rSBA. As pre-specified in protocol, the endpoint was assessed in children and adolescents aged 2 to 17 years in India and RSA as combined groups: Group 5 + Group 7 and Group 6 + Group 8 as they received the same dose of MenACYW conjugate vaccine and Menactra® respectively.
Time Frame: Day 0 (pre-vaccination) and Day 30 (30 days post-vaccination on Day 0)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 5 + Group 7: MenACYW Conjugate Vaccine | Group 6 + Group 8: Menactra®
Number analyzed (Participants) | 445 | 445
titer
  hSBA: Serogroup A: Day 0 | 7.40 [6.79 to 8.07] | 7.21 [6.66 to 7.80]
  hSBA: Serogroup A: Day 30: number analyzed (Participants) | 443 | 443
  hSBA: Serogroup A: Day 30 | 56.1 [48.5 to 65.0] | 36.3 [31.0 to 42.5]
  hSBA: Serogroup C: Day 0 | 3.97 [3.63 to 4.34] | 3.78 [3.46 to 4.13]
  hSBA: Serogroup C: Day 30: number analyzed (Participants) | 445 | 443
  hSBA: Serogroup C: Day 30 | 600 [521 to 692] | 47.3 [38.3 to 58.4]
  hSBA: Serogroup Y: Day 0: number analyzed (Participants) | 443 | 445
  hSBA: Serogroup Y: Day 0 | 3.50 [3.13 to 3.91] | 3.50 [3.14 to 3.91]
  hSBA: Serogroup Y: Day 30: number analyzed (Participants) | 445 | 443
  hSBA: Serogroup Y: Day 30 | 167 [145 to 191] | 46.2 [39.3 to 54.3]
  hSBA: Serogroup W: Day 0 | 4.31 [3.88 to 4.78] | 4.04 [3.65 to 4.48]
  hSBA: Serogroup W: Day 30 | 121 [106 to 137] | 35.4 [30.4 to 41.1]
  rSBA: Serogroup A: Day 0: number analyzed (Participants) | 186 | 189
  rSBA: Serogroup A: Day 0 | 308 [199 to 478] | 387 [260 to 577]
  rSBA: Serogroup A: Day 30: number analyzed (Participants) | 191 | 189
  rSBA: Serogroup A: Day 30 | 10561 [9223 to 12094] | 8313 [7275 to 9499]
  rSBA: Serogroup C: Day 0: number analyzed (Participants) | 191 | 190
  rSBA: Serogroup C: Day 0 | 3.56 [2.91 to 4.36] | 3.73 [3.02 to 4.62]
  rSBA: Serogroup C: Day 30: number analyzed (Participants) | 191 | 189
  rSBA: Serogroup C: Day 30 | 14430 [11923 to 17463] | 1199 [869 to 1655]
  rSBA: Serogroup Y: Day 0: number analyzed (Participants) | 181 | 182
  rSBA: Serogroup Y: Day 0 | 17.3 [11.5 to 26.2] | 21.9 [14.4 to 33.4]
  rSBA: Serogroup Y: Day 30: number analyzed (Participants) | 191 | 188
  rSBA: Serogroup Y: Day 30 | 15404 [13409 to 17696] | 5966 [4850 to 7339]
  rSBA: Serogroup W: Day 0: number analyzed (Participants) | 189 | 189
  rSBA: Serogroup W: Day 0 | 7.01 [5.00 to 9.83] | 7.46 [5.36 to 10.4]
  rSBA: Serogroup W: Day 30: number analyzed (Participants) | 191 | 189
  rSBA: Serogroup W: Day 30 | 19644 [16338 to 23618] | 6598 [5160 to 8437]

7. Secondary Outcome: Group 5 and Group 6: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured by hSBA and rSBA.
Time Frame: Day 0 (pre-vaccination) and Day 30 (30 days post-vaccination on Day 0)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 5: MenACYW Conjugate Vaccine | Group 6: Menactra®
Number analyzed (Participants) | 222 | 228
titer
  hSBA: Serogroup A: Day 0 | 7.33 [6.50 to 8.26] | 7.71 [6.94 to 8.58]
  hSBA: Serogroup A: Day 30: number analyzed (Participants) | 220 | 228
  hSBA: Serogroup A: Day 30 | 70.3 [56.5 to 87.6] | 40.9 [32.8 to 51.1]
  hSBA: Serogroup C: Day 0 | 3.36 [3.00 to 3.76] | 3.17 [2.84 to 3.55]
  hSBA: Serogroup C: Day 30 | 595 [494 to 716] | 38.3 [28.4 to 51.6]
  hSBA: Serogroup Y: Day 0 | 3.32 [2.84 to 3.88] | 3.12 [2.70 to 3.60]
  hSBA: Serogroup Y: Day 30 | 119 [97.4 to 145] | 27.1 [21.7 to 33.8]
  hSBA: Serogroup W: Day 0 | 3.23 [2.86 to 3.65] | 2.85 [2.56 to 3.17]
  hSBA: Serogroup W: Day 30 | 92.8 [78.7 to 109] | 24.3 [19.8 to 29.7]
  rSBA: Serogroup A: Day 0: number analyzed (Participants) | 92 | 98
  rSBA: Serogroup A: Day 0 | 159 [81.9 to 310] | 337 [188 to 605]
  rSBA: Serogroup A: Day 30: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup A: Day 30 | 11462 [9425 to 13938] | 6877 [5755 to 8217]
  rSBA: Serogroup C: Day 0: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup C: Day 0 | 3.09 [2.39 to 4.01] | 2.98 [2.40 to 3.70]
  rSBA: Serogroup C: Day 30: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup C: Day 30 | 11139 [8843 to 14030] | 659 [413 to 1052]
  rSBA: Serogroup Y: Day 0: number analyzed (Participants) | 87 | 91
  rSBA: Serogroup Y: Day 0 | 11.4 [6.25 to 20.6] | 18.8 [10.4 to 33.7]
  rSBA: Serogroup Y: Day 30: number analyzed (Participants) | 97 | 98
  rSBA: Serogroup Y: Day 30 | 15696 [12565 to 19609] | 4522 [3316 to 6168]
  rSBA: Serogroup W: Day 0: number analyzed (Participants) | 95 | 98
  rSBA: Serogroup W: Day 0 | 6.62 [4.10 to 10.7] | 7.78 [4.78 to 12.7]
  rSBA: Serogroup W: Day 30: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup W: Day 30 | 19037 [14748 to 24572] | 4332 [2969 to 6320]

8. Secondary Outcome: Group 5 and Group 6: Percentage of Participants Who Achieved Antibody Titers ≥Pre-defined Thresholds Against Meningococcal Serogroups A, C, Y, and W
Description: as for outcome 3
Time Frame: Day 0 (pre-vaccination) and Day 30 (30 days post-vaccination on Day 0)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: MenACYW Conjugate Vaccine | Group 6: Menactra®
Number analyzed (Participants) | 222 | 228
percentage of participants
  hSBA: Serogroup A: Day 0: ≥1:4 | 85.1 [79.8 to 89.5] | 91.2 [86.8 to 94.6]
  hSBA: Serogroup A: Day 0: ≥1:8 | 60.8 [54.1 to 67.3] | 63.6 [57.0 to 69.8]
  hSBA: Serogroup A: Day 30: ≥1:4: number analyzed (Participants) | 220 | 228
  hSBA: Serogroup A: Day 30: ≥1:4 | 92.3 [87.9 to 95.4] | 94.7 [91.0 to 97.3]
  hSBA: Serogroup A: Day 30: ≥1:8: number analyzed (Participants) | 220 | 228
  hSBA: Serogroup A: Day 30: ≥1:8 | 89.5 [84.7 to 93.3] | 83.8 [78.3 to 88.3]
  hSBA: Serogroup C: Day 0: ≥1:4 | 37.8 [31.4 to 44.6] | 30.7 [24.8 to 37.1]
  hSBA: Serogroup C: Day 0: ≥1:8 | 19.8 [14.8 to 25.7] | 18.4 [13.6 to 24.1]
  hSBA: Serogroup C: Day 30: ≥1:4 | 99.5 [97.5 to 100] | 82.9 [77.4 to 87.5]
  hSBA: Serogroup C: Day 30: ≥1:8 | 99.5 [97.5 to 100] | 72.8 [66.5 to 78.5]
  hSBA: Serogroup Y: Day 0: ≥1:4 | 21.2 [16.0 to 27.1] | 18.9 [14.0 to 24.6]
  hSBA: Serogroup Y: Day 0: ≥1:8 | 16.2 [11.6 to 21.7] | 13.6 [9.4 to 18.7]
  hSBA: Serogroup Y: Day 30: ≥1:4 | 94.1 [90.2 to 96.8] | 83.8 [78.3 to 88.3]
  hSBA: Serogroup Y: Day 30: ≥1:8 | 93.7 [89.6 to 96.5] | 76.8 [70.7 to 82.1]
  hSBA: Serogroup W: Day 0: ≥1:4 | 27.9 [22.1 to 34.3] | 20.2 [15.2 to 26.0]
  hSBA: Serogroup W: Day 0: ≥1:8 | 18.9 [14.0 to 24.7] | 13.6 [9.4 to 18.7]
  hSBA: Serogroup W: Day 30: ≥1:4 | 99.1 [96.8 to 99.9] | 86.8 [81.8 to 90.9]
  hSBA: Serogroup W: Day 30: ≥1:8 | 98.2 [95.5 to 99.5] | 82.0 [76.4 to 86.8]
  rSBA: Serogroup A: Day 0: ≥1:8: number analyzed (Participants) | 92 | 98
  rSBA: Serogroup A: Day 0: ≥1:8 | 66.3 [55.7 to 75.8] | 76.5 [66.9 to 84.5]
  rSBA: Serogroup A: Day 0: ≥1:128: number analyzed (Participants) | 92 | 98
  rSBA: Serogroup A: Day 0: ≥1:128 | 62.0 [51.2 to 71.9] | 73.5 [63.6 to 81.9]
  rSBA: Serogroup A: Day 30: ≥1:8: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup A: Day 30: ≥1:8 | 100 [96.3 to 100] | 100 [96.3 to 100]
  rSBA: Serogroup A: Day 30: ≥1:128: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup A: Day 30: ≥1:128 | 100 [96.3 to 100] | 100 [96.3 to 100]
  rSBA: Serogroup C: Day 0: ≥1:8: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup C: Day 0: ≥1:8 | 11.3 [5.8 to 19.4] | 13.1 [7.2 to 21.4]
  rSBA: Serogroup C: Day 0: ≥1:128: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup C: Day 0: ≥1:128 | 5.2 [1.7 to 11.6] | 4.0 [1.1 to 10.0]
  rSBA: Serogroup C: Day 30: ≥1:8: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup C: Day 30: ≥1:8 | 100 [96.3 to 100] | 90.9 [83.4 to 95.8]
  rSBA: Serogroup C: Day 30: ≥1:128: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup C: Day 30: ≥1:128 | 100 [96.3 to 100] | 85.9 [77.4 to 92.0]
  rSBA: Serogroup Y: Day 0: ≥1:8: number analyzed (Participants) | 87 | 91
  rSBA: Serogroup Y: Day 0: ≥1:8 | 28.7 [19.5 to 39.4] | 40.7 [30.5 to 51.5]
  rSBA: Serogroup Y: Day 0: ≥1:128: number analyzed (Participants) | 87 | 91
  rSBA: Serogroup Y: Day 0: ≥1:128 | 28.7 [19.5 to 39.4] | 38.5 [28.4 to 49.2]
  rSBA: Serogroup Y: Day 30: ≥1:8: number analyzed (Participants) | 97 | 98
  rSBA: Serogroup Y: Day 30: ≥1:8 | 100 [96.3 to 100] | 98.0 [92.8 to 99.8]
  rSBA: Serogroup Y: Day 30: ≥1:128: number analyzed (Participants) | 97 | 98
  rSBA: Serogroup Y: Day 30: ≥1:128 | 100 [96.3 to 100] | 98.0 [92.8 to 99.8]
  rSBA: Serogroup W: Day 0: ≥1:8: number analyzed (Participants) | 95 | 98
  rSBA: Serogroup W: Day 0: ≥1:8 | 21.1 [13.4 to 30.6] | 24.5 [16.4 to 34.2]
  rSBA: Serogroup W: Day 0: ≥1:128: number analyzed (Participants) | 95 | 98
  rSBA: Serogroup W: Day 0: ≥1:128 | 21.1 [13.4 to 30.6] | 24.5 [16.4 to 34.2]
  rSBA: Serogroup W: Day 30: ≥1:8: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup W: Day 30: ≥1:8 | 100 [96.3 to 100] | 98.0 [92.9 to 99.8]
  rSBA: Serogroup W: Day 30: ≥1:128: number analyzed (Participants) | 97 | 99
  rSBA: Serogroup W: Day 30: ≥1:128 | 100 [96.3 to 100] | 97.0 [91.4 to 99.4]

9. Secondary Outcome: Group 7 and Group 8: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured by hSBA and rSBA.
Time Frame: Day 0 (pre-vaccination) and Day 30 (30 days post-vaccination on Day 0)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 7: MenACYW Conjugate Vaccine | Group 8: Menactra®
Number analyzed (Participants) | 223 | 217
titer
  hSBA: Serogroup A: Day 0 | 7.47 [6.59 to 8.47] | 6.71 [5.97 to 7.55]
  hSBA: Serogroup A: Day 30: number analyzed (Participants) | 223 | 215
  hSBA: Serogroup A: Day 30 | 44.9 [37.1 to 54.4] | 31.9 [25.5 to 40.0]
  hSBA: Serogroup C: Day 0 | 4.69 [4.10 to 5.36] | 4.55 [3.97 to 5.20]
  hSBA: Serogroup C: Day 30: number analyzed (Participants) | 223 | 215
  hSBA: Serogroup C: Day 30 | 606 [488 to 751] | 59.2 [44.0 to 79.7]
  hSBA: Serogroup Y: Day 0: number analyzed (Participants) | 221 | 217
  hSBA: Serogroup Y: Day 0 | 3.69 [3.13 to 4.34] | 3.96 [3.35 to 4.69]
  hSBA: Serogroup Y: Day 30: number analyzed (Participants) | 223 | 215
  hSBA: Serogroup Y: Day 30 | 233 [195 to 279] | 81.5 [66.0 to 101]
  hSBA: Serogroup W: Day 0 | 5.74 [4.89 to 6.74] | 5.85 [4.97 to 6.88]
  hSBA: Serogroup W: Day 30 | 157 [129 to 191] | 52.5 [42.3 to 65.2]
  rSBA: Serogroup A: Day 0: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup A: Day 0 | 589 [338 to 1026] | 450 [260 to 778]
  rSBA: Serogroup A: Day 30: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup A: Day 30 | 9706 [8032 to 11729] | 10242 [8432 to 12440]
  rSBA: Serogroup C: Day 0: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup C: Day 0 | 4.12 [3.00 to 5.66] | 4.77 [3.28 to 6.93]
  rSBA: Serogroup C: Day 30: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup C: Day 30 | 18848 [13953 to 25460] | 2317 [1544 to 3476]
  rSBA: Serogroup Y: Day 0: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup Y: Day 0 | 25.6 [14.6 to 45.2] | 25.7 [13.9 to 47.3]
  rSBA: Serogroup Y: Day 30: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup Y: Day 30 | 15108 [12775 to 17865] | 8067 [6207 to 10483]
  rSBA: Serogroup W: Day 0: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup W: Day 0 | 7.43 [4.57 to 12.1] | 7.14 [4.55 to 11.2]
  rSBA: Serogroup W: Day 30: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup W: Day 30 | 20290 [15479 to 26598] | 10481 [7890 to 13924]

10. Secondary Outcome: Group 7 and Group 8: Percentage of Participants Who Achieved Antibody Titers ≥Pre-defined Thresholds Against Meningococcal Serogroups A, C, Y, and W
Description: as for outcome 3
Time Frame: Day 0 (pre-vaccination) and Day 30 (30 days post-vaccination on Day 0)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 7: MenACYW Conjugate Vaccine | Group 8: Menactra®
Number analyzed (Participants) | 223 | 217
percentage of participants
  hSBA: Serogroup A: Day 0: ≥1:4 | 88.8 [83.9 to 92.6] | 86.6 [81.4 to 90.9]
  hSBA: Serogroup A: Day 0: ≥1:8 | 61.0 [54.2 to 67.4] | 57.6 [50.7 to 64.3]
  hSBA: Serogroup A: Day 30: ≥1:4: number analyzed (Participants) | 223 | 215
  hSBA: Serogroup A: Day 30: ≥1:4 | 96.9 [93.6 to 98.7] | 93.5 [89.3 to 96.4]
  hSBA: Serogroup A: Day 30: ≥1:8: number analyzed (Participants) | 223 | 215
  hSBA: Serogroup A: Day 30: ≥1:8 | 89.7 [84.9 to 93.3] | 82.3 [76.6 to 87.2]
  hSBA: Serogroup C: Day 0: ≥1:4 | 58.3 [51.5 to 64.8] | 57.1 [50.3 to 63.8]
  hSBA: Serogroup C: Day 0: ≥1:8 | 32.3 [26.2 to 38.9] | 30.4 [24.4 to 37.0]
  hSBA: Serogroup C: Day 30: ≥1:4: number analyzed (Participants) | 223 | 215
  hSBA: Serogroup C: Day 30: ≥1:4 | 99.6 [97.5 to 100] | 93.0 [88.8 to 96.0]
  hSBA: Serogroup C: Day 30: ≥1:8: number analyzed (Participants) | 223 | 215
  hSBA: Serogroup C: Day 30: ≥1:8 | 99.1 [96.8 to 99.9] | 82.8 [77.1 to 87.6]
  hSBA: Serogroup Y: Day 0: ≥1:4: number analyzed (Participants) | 221 | 217
  hSBA: Serogroup Y: Day 0: ≥1:4 | 28.1 [22.2 to 34.5] | 32.3 [26.1 to 38.9]
  hSBA: Serogroup Y: Day 0: ≥1:8: number analyzed (Participants) | 221 | 217
  hSBA: Serogroup Y: Day 0: ≥1:8 | 21.3 [16.1 to 27.3] | 25.3 [19.7 to 31.7]
  hSBA: Serogroup Y: Day 30: ≥1:4: number analyzed (Participants) | 223 | 215
  hSBA: Serogroup Y: Day 30: ≥1:4 | 99.6 [97.5 to 100] | 95.8 [92.2 to 98.1]
  hSBA: Serogroup Y: Day 30: ≥1:8: number analyzed (Participants) | 223 | 215
  hSBA: Serogroup Y: Day 30: ≥1:8 | 99.6 [97.5 to 100] | 94.9 [91.0 to 97.4]
  hSBA: Serogroup W: Day 0: ≥1:4 | 53.4 [46.6 to 60.1] | 55.3 [48.4 to 62.0]
  hSBA: Serogroup W: Day 0: ≥1:8 | 42.2 [35.6 to 48.9] | 41.0 [34.4 to 47.9]
  hSBA: Serogroup W: Day 30: ≥1:4 | 99.1 [96.8 to 99.9] | 94.9 [91.1 to 97.4]
  hSBA: Serogroup W: Day 30: ≥1:8 | 99.1 [96.8 to 99.9] | 93.5 [89.4 to 96.4]
  rSBA: Serogroup A: Day 0: ≥1:8: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup A: Day 0: ≥1:8 | 84.0 [75.0 to 90.8] | 83.5 [74.3 to 90.5]
  rSBA: Serogroup A: Day 0: ≥1:128: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup A: Day 0: ≥1:128 | 81.9 [72.6 to 89.1] | 80.2 [70.6 to 87.8]
  rSBA: Serogroup A: Day 30: ≥1:8: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup A: Day 30: ≥1:8 | 100 [96.2 to 100] | 100 [96.0 to 100]
  rSBA: Serogroup A: Day 30: ≥1:128: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup A: Day 30: ≥1:128 | 100 [96.2 to 100] | 100 [96.0 to 100]
  rSBA: Serogroup C: Day 0: ≥1:8: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup C: Day 0: ≥1:8 | 19.1 [11.8 to 28.6] | 19.8 [12.2 to 29.4]
  rSBA: Serogroup C: Day 0: ≥1:128: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup C: Day 0: ≥1:128 | 6.4 [2.4 to 13.4] | 9.9 [4.6 to 17.9]
  rSBA: Serogroup C: Day 30: ≥1:8: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup C: Day 30: ≥1:8 | 100 [96.2 to 100] | 98.9 [94.0 to 100]
  rSBA: Serogroup C: Day 30: ≥1:128: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup C: Day 30: ≥1:128 | 100 [96.2 to 100] | 96.7 [90.6 to 99.3]
  rSBA: Serogroup Y: Day 0: ≥1:8: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup Y: Day 0: ≥1:8 | 47.9 [37.5 to 58.4] | 46.2 [35.6 to 56.9]
  rSBA: Serogroup Y: Day 0: ≥1:128: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup Y: Day 0: ≥1:128 | 46.8 [36.4 to 57.4] | 40.7 [30.5 to 51.5]
  rSBA: Serogroup Y: Day 30: ≥1:8: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup Y: Day 30: ≥1:8 | 100 [96.2 to 100] | 98.9 [94.0 to 100]
  rSBA: Serogroup Y: Day 30: ≥1:128: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup Y: Day 30: ≥1:128 | 100 [96.2 to 100] | 98.9 [94.0 to 100]
  rSBA: Serogroup W: Day 0: ≥1:8: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup W: Day 0: ≥1:8 | 24.5 [16.2 to 34.4] | 26.4 [17.7 to 36.7]
  rSBA: Serogroup W: Day 0: ≥1:128: number analyzed (Participants) | 94 | 91
  rSBA: Serogroup W: Day 0: ≥1:128 | 22.3 [14.4 to 32.1] | 23.1 [14.9 to 33.1]
  rSBA: Serogroup W: Day 30: ≥1:8: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup W: Day 30: ≥1:8 | 100 [96.2 to 100] | 100 [96.0 to 100]
  rSBA: Serogroup W: Day 30: ≥1:128: number analyzed (Participants) | 94 | 90
  rSBA: Serogroup W: Day 30: ≥1:128 | 100 [96.2 to 100] | 100 [96.0 to 100]

ADVERSE EVENTS:
Time Frame: From the first study vaccine administration (Day 0) up to 30 days post-vaccination on Day 0, mean study subject duration was 33 days for Groups 1 to 4, 34 days for Groups 5 and 6, and 35 days for Groups 7 and 8.
Description: Analysis was performed on safety analysis set which was defined as those participants who received at least 1 dose of the study vaccine and had any safety data available. All participants had their safety analyzed according to the vaccine they actually received.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® | Group 3: MenACYW Conjugate Vaccine | Group 4: Quadri Meningo™/Locally Available Licensed Meningococcal Vaccine | Group 5: MenACYW Conjugate Vaccine | Group 6: Menactra® | Group 7: MenACYW Conjugate Vaccine | Group 8: Menactra®
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/100 | 0/100 | 0/100 | 0/232 | 0/232 | 0/229 | 0/227
Serious Adverse Events (participants affected / at risk) | 1/98 | 0/100 | 0/100 | 0/100 | 1/232 | 0/232 | 0/229 | 0/227
Other Adverse Events (participants affected / at risk) | 32/98 | 26/100 | 18/100 | 21/100 | 81/232 | 43/232 | 115/229 | 128/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=98) | Group 2: Menactra® (N=100) | Group 3: MenACYW Conjugate Vaccine (N=100) | Group 4: Quadri Meningo™/Locally Available Licensed Meningococcal Vaccine (N=100) | Group 5: MenACYW Conjugate Vaccine (N=232) | Group 6: Menactra® (N=232) | Group 7: MenACYW Conjugate Vaccine (N=229) | Group 8: Menactra® (N=227)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue Fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=98) | Group 2: Menactra® (N=100) | Group 3: MenACYW Conjugate Vaccine (N=100) | Group 4: Quadri Meningo™/Locally Available Licensed Meningococcal Vaccine (N=100) | Group 5: MenACYW Conjugate Vaccine (N=232) | Group 6: Menactra® (N=232) | Group 7: MenACYW Conjugate Vaccine (N=229) | Group 8: Menactra® (N=227)
Injection Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 28 (28) | 27 (27)
Injection Site Pain (General disorders) | 27 (27) | 24 (24) | 9 (9) | 14 (14) | 52 (52) | 29 (29) | 85 (85) | 82 (82)
Injection Site Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 25 (25) | 37 (37)
Malaise (General disorders) | 6 (6) | 5 (5) | 1 (1) | 1 (1) | 11 (11) | 4 (4) | 45 (45) | 44 (44)
Pyrexia (General disorders) | 5 (5) | 2 (2) | 4 (4) | 4 (4) | 37 (37) | 16 (16) | 8 (8) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 2 (2) | 0 (0) | 7 (7) | 3 (3) | 46 (46) | 49 (49)
Headache (Nervous system disorders) | 6 (6) | 6 (6) | 3 (3) | 3 (3) | 13 (13) | 3 (3) | 56 (57) | 57 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT04143061/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT04143061/SAP_001.pdf